CLINICAL TRIAL: NCT06209788
Title: The Efficacy of Music in Preventing Delirium in Elderly Patients With Hip Fracture: A Randomized Controlled Trial
Brief Title: The Efficacy of Music in Preventing Delirium in Elderly Patients With Hip Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Han-Chang Ku, PhD & Assistant Professor, RN, Chang Gung University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CYCH2023084
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Delirium in Old Age; Hip Fractures
Keywords: delirium; hip fracture; music; randomized controlled trial
MeSH Terms: conditions — Hip Fractures; Delirium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The music intervention consists of two parts. The first part occurs during the surgical procedure, starting from the induction of anesthesia and continuing until the surgery over. The second part spans from the first day post-surgery to the fifth day (or until discharge), with the patient listening to music twice a day, each session lasting for 30 minutes. The planned times for the music sessions are expected to be at 11 a.m. and 8 p.m. Each day post-surgery, the music intervention must be completed, and measurements of respiratory rate, pulse rate, blood pressure, and pain score should be taken both before and after listening to the music. Other are routine post-operative care.
  Interventions: Procedure: experimental group
- Control group (No Intervention): Routine post-operative care.

INTERVENTIONS:
Procedure: experimental group — The music intervention consists of two parts. The first part occurs during the surgical procedure, starting from the induction of anesthesia and continuing until the surgery over. The second part spans from the first day post-surgery to the fifth day (or until discharge), with the patient listening to music twice a day, each session lasting for 30 minutes. The planned times for the music sessions are expected to be at 11 a.m. and 8 p.m. Each day post-surgery, the music intervention must be completed, and measurements of respiratory rate, pulse rate, blood pressure, and pain score should be taken both before and after listening to the music. Other are routine post-operative care.
  Arms: Experimental group

SUMMARY:
The aim of this trial is to explore the efficacy of music in preventing delirium in elderly patients with hip fracture.

The main aims of this research are:

1. To compare the effectiveness of music intervention in preventing delirium in patients with hip fractures through a randomized controlled trial. The comparisons include respiratory rate, pulse rate, blood pressure, and pain score, as well as the incidence and severity of delirium, opioid analgesic usage, postoperative complications, length of hospital stay, and rates of readmission within 14 days and 30-day mortality.
2. Introduce the evidence-based ''listening music protocol'' in the care of hip fracture patients to prevent delirium, and test the effects through a randomized controlled trial.

DETAILED DESCRIPTION:
This study is a two-group, pre and post-test, randomized controlled trial to test the effectiveness of the ''listening music protocol''. Convenience sampling will be used to select the inpatients with hip fractures in a regional hospital in southern Taiwan. 102 participants will be randomly assigned either to an experimental (n=51) or to a control (n=51) group. The experimental group will receive a six-day music protocol and regular post-operative care. The control group will receive regular post-operative care only. Statistical analysis was performed using SPSS Version 22.0.

Descriptive statistics, including frequencies, percentages, means, and medians, were used to analyze basic attributes. For the analysis of homogeneity, the chi-square test or Fisher's exact test was employed for categorical variables. The paired t-test was used to compare respiratory rate, pulse rate, blood pressure, and pain index.

Following the intervention, the occurrence and severity of delirium before and after implementing music intervention were compared. Additionally, comparisons were made for opioid analgesic usage, postoperative complications, length of hospital stay, and 30-day mortality.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 65 years and above (inclusive).
* Individuals with clear consciousness and willingness to participate in this study.
* The primary treating physician of the participant must be the principal investigator or co-principal investigator of this study.
* Diagnosis of femoral head fracture, femoral neck fracture, or intertrochanteric fracture.
* Surgical procedures include hip hemiarthroplasty, total hip arthroplasty, cannulated screw fixation, dynamic hip screw, femoral neck system, and gamma-nail.

Exclusion Criteria:

* Bilateral hip fractures simultaneously.
* History of neurosurgery.
* Preoperative delirium.
* Severe hearing impairment (unable to engage in oral conversation).
* Use of sedatives or antidepressant medications.
* Dementia or psychiatric disorders.
* Patient unwilling to participate in the study or cooperate with listening to music (using headphones).
* Use of unknown medications and alcohol.
* After taking antihypertensive medication, preoperative systolic blood pressure >200 mmHg or diastolic blood pressure >110 mmHg.
* Preoperative heart rate >130 beats per minute or <50 beats per minute.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-01-15 (Estimated); Primary Completion 2024-12-05 (Estimated); Study Completion 2024-12-05 (Estimated)

PRIMARY OUTCOMES:
delirium event and severity | 7-14 days
  Delirium is diagnosed based on clinical symptoms, utilizing the Confusion Assessment Method (CAM) to assess. CAM consists of four elements that can be quickly completed in a hospital setting, making it a convenient diagnostic tool. The four components include abrupt onset, fluctuating course of symptoms, inattention, and disorganized thinking or altered level of consciousness.

SECONDARY OUTCOMES:
opioid analgesic usage | 7-14 days
  Comparison of patients' opioid analgesic dosage and frequency during hospitalization.
postoperative complications | 1 month
  Comparison of surgical complications occurring during hospitalization or within one month post-discharge.
length of hospital stay | 7-14 days
  Comparison of patients' length of hospital stay during hospitalization.
readmission within 14 days postoperatively | 1 month
  Recording whether patients are readmitted within 14 days post-discharge due to surgical complications or delirium.
30-day mortality | 1 month
  Recording whether patients die within 30 days post-discharge due to surgical complications or delirium issues.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] American Geriatrics Society Expert Panel on Postoperative Delirium in Older Adults. Postoperative delirium in older adults: best practice statement from the American Geriatrics Society. J Am Coll Surg. 2015 Feb;220(2):136-48.e1. doi: 10.1016/j.jamcollsurg.2014.10.019. Epub 2014 Nov 14. No abstract available. PMID 25535170
- [Result] Chen Y, Liang S, Wu H, Deng S, Wang F, Lunzhu C, Li J. Postoperative delirium in geriatric patients with hip fractures. Front Aging Neurosci. 2022 Dec 22;14:1068278. doi: 10.3389/fnagi.2022.1068278. eCollection 2022. PMID 36620772
- [Result] Chlan LL, Weinert CR, Heiderscheit A, Tracy MF, Skaar DJ, Guttormson JL, Savik K. Effects of patient-directed music intervention on anxiety and sedative exposure in critically ill patients receiving mechanical ventilatory support: a randomized clinical trial. JAMA. 2013 Jun 12;309(22):2335-44. doi: 10.1001/jama.2013.5670. PMID 23689789
- [Result] Esfahanian F, Mirmohammadsadeghi A, Gholami H, Neshat S, Mansouri M, Sadeghi M, Bathaie SR, Heidari Z, Mirmohammadsadeghi M. Using Music for the Prevention of Delirium in Patients After Coronary Artery Bypass Graft Surgery: A Randomized Clinical Trial. J Cardiothorac Vasc Anesth. 2022 Dec;36(12):4341-4346. doi: 10.1053/j.jvca.2022.09.007. Epub 2022 Sep 9. PMID 36241502
- [Result] Fu VX, Jeekel J, Van Lieshout EMM, Van der Velde D, Slegers LJP, Haverlag R, Haumann J, Poley MJ, Verhofstad MHJ; MCHOPIN collaborators. Effect of music on clinical outcome after hip fracture operations (MCHOPIN): study protocol of a multicentre randomised controlled trial. BMJ Open. 2021 Dec 23;11(12):e049706. doi: 10.1136/bmjopen-2021-049706. PMID 34949611
- [Result] Golubovic J, Neerland BE, Aune D, Baker FA. Music Interventions and Delirium in Adults: A Systematic Literature Review and Meta-Analysis. Brain Sci. 2022 Apr 28;12(5):568. doi: 10.3390/brainsci12050568. PMID 35624955
- [Result] Haynes MS, Alder KD, Toombs C, Amakiri IC, Rubin LE, Grauer JN. Predictors and Sequelae of Postoperative Delirium in a Geriatric Patient Population With Hip Fracture. J Am Acad Orthop Surg Glob Res Rev. 2021 May 14;5(5):e20.00221. doi: 10.5435/JAAOSGlobal-D-20-00221. PMID 33989253
- [Result] Igwe EO, Nealon J, Mohammed M, Hickey B, Chou KR, Chen KH, Traynor V. Multi-disciplinary and pharmacological interventions to reduce post-operative delirium in elderly patients: A systematic review and meta-analysis. J Clin Anesth. 2020 Dec;67:110004. doi: 10.1016/j.jclinane.2020.110004. Epub 2020 Aug 5. PMID 32768990
- [Result] Johnson K, Fleury J, McClain D. Music intervention to prevent delirium among older patients admitted to a trauma intensive care unit and a trauma orthopaedic unit. Intensive Crit Care Nurs. 2018 Aug;47:7-14. doi: 10.1016/j.iccn.2018.03.007. Epub 2018 May 4. PMID 29735284
- [Result] Kang J, Cho YS, Lee M, Yun S, Jeong YJ, Won YH, Hong J, Kim S. Effects of nonpharmacological interventions on sleep improvement and delirium prevention in critically ill patients: A systematic review and meta-analysis. Aust Crit Care. 2023 Jul;36(4):640-649. doi: 10.1016/j.aucc.2022.04.006. Epub 2022 Jun 17. PMID 35718628
- [Result] Oh ES, Fong TG, Hshieh TT, Inouye SK. Delirium in Older Persons: Advances in Diagnosis and Treatment. JAMA. 2017 Sep 26;318(12):1161-1174. doi: 10.1001/jama.2017.12067. PMID 28973626
- [Result] Qi YM, Li YJ, Zou JH, Qiu XD, Sun J, Rui YF. Risk factors for postoperative delirium in geriatric patients with hip fracture: A systematic review and meta-analysis. Front Aging Neurosci. 2022 Aug 3;14:960364. doi: 10.3389/fnagi.2022.960364. eCollection 2022. PMID 35992597
- [Result] Ravi B, Pincus D, Choi S, Jenkinson R, Wasserstein DN, Redelmeier DA. Association of Duration of Surgery With Postoperative Delirium Among Patients Receiving Hip Fracture Repair. JAMA Netw Open. 2019 Feb 1;2(2):e190111. doi: 10.1001/jamanetworkopen.2019.0111. PMID 30794305
- [Result] Shin JE, Kyeong S, Lee JS, Park JY, Lee WS, Kim JJ, Yang KH. A personality trait contributes to the occurrence of postoperative delirium: a prospective study. BMC Psychiatry. 2016 Nov 3;16(1):371. doi: 10.1186/s12888-016-1079-z. PMID 27809817
- [Result] Wu J, Yin Y, Jin M, Li B. The risk factors for postoperative delirium in adult patients after hip fracture surgery: a systematic review and meta-analysis. Int J Geriatr Psychiatry. 2021 Jan;36(1):3-14. doi: 10.1002/gps.5408. Epub 2020 Oct 29. PMID 32833302
- [Derived] Chao LY, Lin CC, Wang L, Lu HJ, Chen JL, Ku HC. Effect of music listening on delirium after hip fracture operations (MLDHFO) in a regional hospital in Taiwan: a randomised controlled trial protocol. BMJ Open. 2025 Aug 6;15(8):e095492. doi: 10.1136/bmjopen-2024-095492. PMID 40774707